CLINICAL TRIAL: NCT07054125
Title: The COMPASS Program: Continuous Monitoring, Peer And Structured Support for Management of Uncontrolled Type 2 Diabetes - A Prospective Single-Arm Study
Brief Title: Continuous Glucose Monitoring, Diabetes Education, and Peer Support for Management of Uncontrolled Type 2 Diabetes
Acronym: COMPASS
Status: Recruiting | Type: Observational
Sponsor: Whole Endo (Industry)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 43318527
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus - Poor Control
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Education, lifestyle counseling, and peer support — This research study is investigating whether a diabetes virtual group visit program using a continuous glucose monitor (CGM) can help improve glucose levels and quality of life in individuals with uncontrolled type 2 diabetes.
  People in the study will join group visits virtually to discuss using CGM, understanding CGM, and other information about ways to bring blood sugars to your goal (nutrition, movement, reducing stress, and techniques to start a new habit).

SUMMARY:
This research study is investigating whether a diabetes virtual group visit program using a continuous glucose monitor (CGM) can help improve glucose levels and quality of life in individuals with uncontrolled type 2 diabetes. People in the study will join group visits virtually to discuss using CGM, understanding CGM, and other information about ways to bring blood sugars to your goal (nutrition, movement, reducing stress, and techniques to start a new habit).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosed with type 2 diabetes mellitus Hemoglobin A1c >8% Must have smartphone to connect with continuous glucose monitor

Exclusion Criteria:

* Pregnancy Use of steroids Active cancer treatment Terminal illness Dementia, mental impairment Type 1 diabetes End stage renal disease, on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: North and South Carolina
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Whole Endo, Asheville, North Carolina, United States